CLINICAL TRIAL: NCT04950400
Title: A Study of Camrelizumab Combined With Chemotherapy Sequential Camrelizumab Combined With Apatinib For First-line Treatment of Advanced Non-small Cell Lung Cancer (NSCLC)
Brief Title: A Study of Camrelizumab Combined With Chemotherapy Sequential Camrelizumab Combined With Apatinib Treatment of Advanced NSCLC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Chest Hospital (Other)
Responsible Party: Principal Investigator, Ying Hu, Vice Director, Department of oncology, Beijing Chest Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BJCH-NSCLC-IIT
Record Dates: First submitted 2021-06-29; First posted 2021-07-06 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2021-06

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — camrelizumab; Drug Therapy; apatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Carrelizumab + chemotherapy + apatinib (Experimental)
  Interventions: Drug: Carrelizumab + chemotherapy + apatinib

INTERVENTIONS:
Drug: Carrelizumab + chemotherapy + apatinib — Subjects will receive 200 mg of karizumab every three weeks，Pemetrexed 500 mg / m2 was given on the first day of each cycle,Every three weeks was a period of administration,Carboplatin AUC 5 was given on the first day of each cycle and every three weeks was a cycle，Paclitaxel 175 mg / m2 was given on the first day of each cycle, and every three weeks was an administration cycle，with intravenous drip，Apatinib, 250 mg, oral, once a day (PO, QD), every 3 weeks as a cycle.

SUMMARY:
The purpose of the study is to evaluate the safety and efficacy of camrelizumab combined with chemotherapy in the first-line treatment of advanced in NSCLC patients.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects were 18-70 years old when they signed the informed consent form, and the age was unlimited for men and women;
2. The late stage (Ⅲ b/ Ⅲ C) and stage IV non-small cell lung cancer (according to AICC Eighth Edition) which can not be removed by operation and can not be treated with radical radiotherapy and chemotherapy confirmed by histopathology or cytology;
3. EGFR mutation and alk translocation status were confirmed to be negative at any time after the initial diagnosis;
4. Subjects had not received systemic systemic chemotherapy for advanced / metastatic NSCLC. Chemotherapy and / or radiotherapy are allowed to be used as part of new adjuvant / adjuvant treatment, provided that the treatment has been completed for at least six months before the diagnosis of advanced or metastatic diseases;
5. ECoG score; 0-1 point;
6. According to RECIST v1.1, subjects must have measurable target lesions through CT or MRI examination. The imaging assessment of tumor was performed within 28 days before the first drug use;
7. The main organs function normally, and the test results during screening must meet the following requirements:

1) The blood routine examination standard should meet the requirements (no blood transfusion and blood products within 14 days, no correction by G-CSF and other hematopoietic stimulating factors): A. Hemoglobin (HB) ≥ 90 g/l; B. Neutrophil number (ANC) ≥ 1.5 × 109/L； C. Platelet count (PLT) ≥ 100 × 109/L； 2) Biochemical examination shall meet the following standards: A. TBIL was lower than 1.5 upper limit of normal value (ULN); B. ALT and AST were less than 2.5 ulin, but < 5 uld in liver metastasis; C. The serum creatinine (CR) < 1.5 ULN or the clearance rate of endogenous creatinine was more than 60ml / min (Cockcroft Gault formula); D. The results of routine urine test showed that uro was less than 2+ or 24 hours urinary protein was less than 1G; 8. Men and women of gestational age must agree to take adequate contraceptive measures throughout the study period and within 6 months after the treatment.

Sign written informed consent, and it is expected to be in good compliance with the research plan.

Exclusion Criteria:

1. Mixed NSCLC confirmed by histology or cytology, including mixed squamous cell carcinoma and small cell lung cancer;
2. Previously received anti-PD-1 antibody, anti-PD-L1 antibody, anti-PD-L2 antibody, anti-CTLA-4 antibody (or any other antibody acting on T cell costimulation or checkpoint pathway) or any VEGF / VEGFR inhibitor;
3. Patients with active brain metastases (for patients with stable symptoms of brain metastases after treatment, they can be selected if they remain stable for at least 4 weeks);
4. Imaging evidence of tumor cavity, tumor surrounding or invasion of large blood vessels. In addition, the degree of proximity of the tumor to the large vessels should be considered（ The major vessels in the chest include the main pulmonary artery, left pulmonary artery, right pulmonary artery, four pulmonary veins, superior vena cava, inferior vena cava and aorta.
5. Immunosuppressive drugs were used within 28 days before the first use of karelizumab, excluding nasal and inhaled corticosteroids or physiological doses of systemic steroids (i.e. not more than 10 mg / day prednisolone or other corticosteroids with the same physiological dose of drugs);
6. Received systemic treatment of Chinese herbal medicine with anti-tumor indications or immunomodulatory drugs (including thymosin, interferon and interleukin, except for local use for controlling pleural effusion) within 28 weeks before the first administration;
7. Inoculate live attenuated vaccine within 30 days of the first administration or within the expected period of the study（ For the new coronal vaccine vaccinators, whether they can be selected according to the judgment of the researchers)
8. According to the judgment of the researcher, there is uncontrolled pleural effusion, pericardial effusion or ascites, or the patient has received serous cavity effusion drainage for treatment within 4 weeks before treatment.
9. Subjects with severe infection within 1 month before enrollment, including but not limited to infection complications, bacteremia, severe pneumonia, etc; Subjects with any active infection, or fever of unknown origin > 38.5 ℃ occurred during screening or before the first administration;
10. Patients with active autoimmune disease or immunodeficiency, or with the above-mentioned history, including but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, rheumatoid arthritis, inflammatory bowel disease, hypophysitis, vasculitis, nephritis, etc.) were not included. The following exceptions: Patients with a history of autoimmune hypothyroidism but receiving thyroid hormone replacement therapy were included in the study. After treatment with insulin regimen, patients with type 1 diabetes who have controlled glycemic control can participate in this study.
11. Subjects who received systemic therapy such as bronchodilators were not satisfied with asthma control and could not be included (those who had complete remission of asthma in childhood and did not need any intervention in adulthood could be included).
12. Human immunodeficiency virus (HIV) infection or acquired immune deficiency syndrome (AIDS), untreated active hepatitis B, hepatitis C virus (hepatitis C antibody positive, HCV-RNA higher than the lower limit of analysis method) or co infection of hepatitis B and hepatitis C; Note: the hepatitis B subjects who met the following criteria also met the inclusion criteria: HBV viral load must be <1000 copy /ml (200 IU/ml) before the first dose, and the subjects should be treated with anti HBV therapy during the whole chemotherapy course to avoid virus reactivation. For the subjects with anti HBC (+), HBsAg (-), anti HBS (-) and HBV viral load (-), preventive anti HBV treatment is not necessary, but close monitoring of virus reactivation is needed;
13. Subjects have received or plan to receive solid organ or blood system transplantation (except corneal transplantation) during the study period;
14. Subjects with a history of other malignancies within five years (except for complete treatment of cervical cancer in situ or basal cell carcinoma or squamous cell carcinoma or skin cancer);
15. He has hypertension and cannot be well controlled by antihypertensive drugs (systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg);
16. Clinical symptoms or diseases of heart that can not be well controlled, such as: (1) heart failure of NYHA grade 2 or above; (2) unstable angina pectoris; (3) myocardial infarction within one year; (4) clinically significant supraventricular or ventricular arrhythmia requiring treatment or intervention; (5) QTc > 450ms (male); and; QTc > 470ms (female);
17. Coagulation dysfunction (INR > 2.0, Pt > 16S), bleeding tendency or receiving thrombolytic or anticoagulant therapy, low-dose aspirin and low molecular weight heparin are allowed for prophylactic use;
18. Clinically significant hemoptysis or hemoptysis more than half teaspoon (2.5ml) per day occurred within 2 months before admission; Or significant clinical bleeding symptoms or clear bleeding tendency, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, baseline fecal occult blood + + or above, or vasculitis, etc; There were deep and large ulcers, lesions closely related to big blood vessels and maxilla and mandible;
19. Arteriovenous thrombosis events occurred in the first 6 months, such as cerebrovascular accident (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep venous thrombosis and pulmonary embolism, etc; Known hereditary or acquired bleeding and thrombotic tendency (such as hemophilia, coagulation dysfunction, thrombocytopenia, etc.);
20. Routine urine examination showed that urine protein was ≥ +, and 24-hour urine protein was more than 1.0 G;
21. Currently participating in interventional clinical research treatment, or receiving other experimental drugs or research devices within 4 weeks before the first administration; Not fully recovered from toxicity and / or complications caused by any intervention before the first administration (i.e., ≤ grade 1 or baseline, excluding fatigue or hair loss);
22. Have a clear history of allergy, and may have potential allergy or intolerance to the test drug and its similar biological agents;
23. Those who have a history of psychotropic drug abuse and can not give up or have mental disorders; Other conditions that increase the risk associated with participating in the study or trial drug and, according to the judgment of the investigator, may result in patients not suitable for inclusion in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-07-07 (Estimated); Primary Completion 2023-12-12 (Estimated); Study Completion 2024-04-04 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 1 Year
  From the date Into this study to tumor progression or death for any

SECONDARY OUTCOMES:
Overall survival， | 2 Year
  The time from the beginning of treatment to the death of the subject due to various reasons, calculated by the intended treatment population (ITT)
Objective response rate | 2 Year
  it is defined as the proportion of patients whose tumors shrink to a predetermined size and maintain a minimum time limit. It includes the cases of CR and PR.
Disease Control Rate | 2 Year
  the rate of CR, PR plus SD
Duration of Response | 2 Year
  Cr or PR to the first assessment of PD or death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: ying Hu, doctor, Principal Investigator — Beijing Chest Hospital

IPD SHARING:
Plan to Share IPD: No